CLINICAL TRIAL: NCT05469789
Title: Demographic and Clinical Characteristics, Treatment Patterns, and Real-world Effectiveness of Lanadelumab in Patients With Hereditary Angioedema Type I or II in the United Kingdom: an Ambispective Cohort Study
Brief Title: A Study of Lanadelumab in Teenagers and Adults With Hereditary Angioedema (HAE)
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-0001; MACS-2021-0616012 (Other: Takeda)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug therapy
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prevalent Cohort A: Prevalent Cohort A will comprise eligible participants with HAE type I or II who have initiated treatment with lanadelumab at any point in time (i.e., all prevalent cases of exposure to lanadelumab). The total follow-up encompasses a 12-month pre-treatment period, and an up-to 24-month post-treatment period.
  Interventions: Other: No Intervention
- Prevalent Cohort B: Prevalent Cohort B will comprise eligible participants with HAE type I or II who have been treated with lanadelumab for <12 months (i.e., the subset of participants from Prevalent Cohort A who initiated treatment with lanadelumab within <12 months). The total follow-up encompasses a 12-month pre-treatment and an up to 24-month post-treatment period, as well as a prospective data collection period of participant-specific duration.
  Interventions: Other: No Intervention
- Incident Cohort A: Incident Cohort A will comprise eligible participants with HAE type I or II initiating treatment with lanadelumab at any time within the prospective data collection time period. The total follow-up encompasses a 12-month pre-treatment and an up-to 24-month post-treatment period, as well as a prospective data collection period of participant-specific duration.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As it is an observational study, no intervention is administered in this study.

SUMMARY:
The main aim of this study is to compare the HAE attacks (both total and those requiring on-demand treatment) in the 12 months before and up to 24 months after initiation of treatment with lanadelumab.

This study is conducted in the United Kingdom where participants were treated or about to be treated with landelumab according to their routine practice at hospitals. Data will be directly collected from participants via study diaries, questionnaires, their medical records, and study doctors treating them. Participants will be contacted every 3 months during study participation (via phone).

ELIGIBILITY:
Inclusion:

* Documented diagnosis of HAE type I or II (confirmed through laboratory testing)
* Documented initiation of treatment with lanadelumab or due to be initiated within next 4 weeks
* Greater than or equal to (≥)12 years of age at initiation of treatment with lanadelumab
* ≥12 months of continuous medical record data before initiation of treatment with lanadelumab

Exclusion:

• Exposure to lanadelumab administered as an investigation product in a clinical trial setting at any point in time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey is all participants with HAE type I or II treated with lanadelumab in hospitals within the UK.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Hereditary Angioedema (HAE) Attacks | Up to approximately 3 years
  Number of HAE attacks (both total [including untreated] and those requiring on-demand treatment) will be estimated across the pre- and post-treatment periods (that is, 12 months before and up to 24 months after initiation of treatment with lanadelumab).

SECONDARY OUTCOMES:
Number of Participants Categorized by Their Demographic Characteristics | At index (lanadelumab treatment initiation day)
  Demographic characteristics will include age, sex, and ethnic group at index.
Number of Participants Categorized by Their Clinical Characteristics | Up to approximately 3 years
  Clinical characteristics will include categories of participant-reported age at onset of symptoms, age at diagnosis of HAE, duration of time from onset to diagnosis (i.e., the diagnostic delay), body mass index (BMI) (at index); comorbidities (pre and post index), history of laryngeal attacks (pre index), type of HAE (type I and II), and triggers for HAE symptoms onset (at index and post index). Index is defined as the lanadelumab treatment initiation day.
Number of Participants Categorized by Their Treatment Patterns | At and after index (lanadelumab treatment initiation day plus approximately 2 years)
  Treatment patterns will include categories of the summary of participant-reported duration of lanadelumab treatment, treatment dose given to participants, and participant with switching patterns with lanadelumab on occurence of HAE attacks.
Number of Participants Categorized by Their Patterns of Prophylactic Treatment | Up to approximately 3 years
  Patterns of prophylactic treatment will include categories of the summary of participant-reported use of brand and drug name, duration of treatment, dose of the treatment within same class of prophylactic treatments.
Compare the Number of Participants Categorized by Their Clinical Features of HAE Attacks Before and After Initiation of Lanadelumab | Up to approximately 3 years
  To compare the number clinical features of HAE attacks before and after initiation of lanadelumab. Clinical features of HAE attacks will include categories of summary of participant-reported time of attack, duration of attack, location (e.g., trunk, extremities, and larynx) of HAE attack, the severity (Grade 1 [Mild], Grade 2 [Moderate], and Grade 3 [Severe]) of HAE attack, and hospitalization due to the HAE attack.
Number of Self-Reported HAE Attacks | Up to approximately 3 years
Number of Participants Categorized by Their Clinical Features of Self-Reported HAE Attacks | Up to approximately 3 years
  Clinical features of self-reported HAE attacks will include categories of summary of participant-reported time of attack, duration of attack, location (e.g., trunk, extremities, and larynx) of HAE attack, the severity (Grade 1 [Mild], Grade 2 [Moderate], and Grade 3 [Severe]) of HAE attack, symptoms of HAE attack (e.g., tiredness, abdominal pain, and abdominal swelling), and identified or suspected trigger(s) for the attack (e.g., contact with chemicals, drugs, or foods).
European Quality of Life 5 Dimensions 3-levels (EQ-5D-3L) Questionnaire Total Score | Up to approximately 2 years
  The EQ-5D-5L questionnaire will be used to record impact of HAE on participant's quality-of-life (QoL). The EQ-5D-5L is a descriptive system of Health-Related Quality-of-Life (HRQoL) states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take 1 of 5 responses. The responses record 5 levels of severity [no problems, slight problems, moderate problems, severe problems, and extreme problems] within a particular dimension. The scores will be the sum of scores from each dimension and can range from 5 (no problems) to 25 (extreme problems). Higher score indicated a worsening health condition.
EQ-5D-3L Visual Analogue Scale (VAS) Score | Up to approximately 2 years
  The EQ-5D-3L VAS records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS is used as a quantitative measure of health outcome that reflect the participant's own judgement score, with a score of 0 as the worst and 100 as the best possible health.
Angioedema Quality of Life (AE-QoL) Total Scores | Up to approximately 2 years
  AE-QoL is a self-administered instrument designed to measure HRQoL in adult participants with recurrent angioedema. The AE-QoL consists of 17 disease-specific quality-of-life items, to produce a total AE-QoL score and 4 domain scores (functioning, fatigue/mood, fears/shame, and food, Each of the 17 items has a five-point response scale ranging from 1 (Never) to 5 (Very Often).
Angioedema Quality of Life (AE-QoL) Domain Scores | Up to approximately 2 years
  AE-QoL is a self-administered instrument designed to measure HRQoL in adult participants with recurrent angioedema. The AE-QoL consists of 17 disease-specific quality-of-life items, to produce a total AE-QoL score and 4 domain scores (functioning, fatigue/mood, fears/shame, and food, Each of the 17 items has a five-point response scale ranging from 1 (Never) to 5 (Very Often).
Number of Participants With HAE-related Health Care Resource Utilization (HCRU) | Up to approximately 3 years
  Healthcare resources used during medical encounters include in and out-patient visits to physicians, hospital admissions, in and out-patient emergency care, and in and out-patient clinical examinations and tests.
Angioedema Control Test (AECT) Total Score | Up to approximately 2 years
  The AECT is used to assess participants with recurrent angioedema. The test uses a questionnaire with 4 items, each of which has 5 options and is used to measure the participant's current disease control. HAE control score will be recorded with 5 levels of answers [1=very often, 2=often, 3=sometimes, 4=seldom, 5=not at all] to the following questions: 1) In the last 3 months, how often have you had angioedema? 2) In the last 3 months, how much has your QoL been affected by angioedema? 3) In the last 3 months, how much has the unpredictability of your angioedema bothered you? 4) In the last 3 months, how well has your angioedema been controlled by your therapy?
Angioedema Control Test (AECT) Domain Score | Up to approximately 2 years
  The AECT is used to assess participants with recurrent angioedema. The test uses a questionnaire with 4 items, each of which has 5 options and is used to measure the participant's current disease control. HAE control score will be recorded with 5 levels of answers [1=very often, 2=often, 3=sometimes, 4=seldom, 5=not at all] to the following questions: 1) In the last 3 months, how often have you had angioedema? 2) In the last 3 months, how much has your QoL been affected by angioedema? 3) In the last 3 months, how much has the unpredictability of your angioedema bothered you? 4) In the last 3 months, how well has your angioedema been controlled by your therapy?
Treatment Satisfaction Questionnaire for Medication (TSQM) Total Score | Up to approximately 2 years
  The TSQM comprises 14 items across four domains focusing on effectiveness (three items), side effects (five items), convenience (three items), and global satisfaction (three items) of the medication over the previous 2-3 weeks, or since the patient's last use. With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). The 7-item scales had a non-neutral midpoint, such that there were more positive response options than negative response options, to allow for precise information to be obtained at the upper end of the score distribution. Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100.
Treatment Satisfaction Questionnaire for Medication (TSQM) Domain Score | Up to approximately 2 years
  The TSQM comprises 14 items across four domains focusing on effectiveness (three items), side effects (five items), convenience (three items), and global satisfaction (three items) of the medication over the previous 2-3 weeks, or since the patient's last use. With the exception of item 4 (presence of side effects; yes or no), all items have five or seven responses, scored from one (least satisfied) to five or seven (most satisfied). The 7-item scales had a non-neutral midpoint, such that there were more positive response options than negative response options, to allow for precise information to be obtained at the upper end of the score distribution. Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Barts Health NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/d7c4639cffc94c4e?idFilter=%5B%22TAK-743-0001%22%5D